CLINICAL TRIAL: NCT06520410
Title: Safety and Efficacy of 18 mm Short Vitrectomy Probe for Pediatric Vitreoretinal Surgeries
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 202101643A0
Record Dates: First submitted 2024-02-29; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-02

CONDITIONS: Retinopathy of Prematurity Both Eyes; Retinal Disease; Persistent Fetal Vasculature; Coats Disease; Coats Retinopathy; Familial Exudative Vitreoretinopathies; Vitreous Disorder; Vitreous Anomalies; Retinal Vascular Disorder
MeSH Terms: conditions — Retinal Diseases; Persistent Hyperplastic Primary Vitreous; Retinal Telangiectasis; Familial Exudative Vitreoretinopathies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Short vitrector group (Experimental): All enrolled patients will receive vitrectomy with the 18 mm short vitrectomy probe (25+ Short TOTALPLUS Vit Pak, 7500 CPM, Str Endoillum. w/ RFID, Alcon Laboratories Inc., Fort Worth, TX, USA.) for various vitreoretinopathies.
  Interventions: Device: Pars plana vitrectomy with a 18 mm short vitrector

INTERVENTIONS:
Device: Pars plana vitrectomy with a 18 mm short vitrector — Using the shorter 18 mm vitrector for various pediatric vitreoretinal surgeries

SUMMARY:
This study aims to study the safety and efficacy of using an 18 mm short vitrectomy probe for pediatric vitreoretinal surgeries and to investigate the surgeon's comfort and reliability of using the shorter probe.

DETAILED DESCRIPTION:
With advancements in sutureless vitrectomy, more and more pediatric disease entities can be successfully coped with intraocular surgeries and with fewer complications. However, the pediatric eye is not just "a smaller adult eye", and pediatric vitreoretinal surgery has its unique challenges. Smaller gauge vitrectomy have evolved from 23-, 25- to 27-gauge, which gave surgeons more intraocular stability, but some issues ensue. The 25- and 27-gauge vitrectors are less stiff, which makes eye rotation and manipulation during vitrectomy more difficult. They are also easier to bend. These alterations force surgeons to change how they perform surgery with 20- or 23-gauge vitrectomy kit. For instance, surgeons have to rely on assistants to do scleral indentation to view the periphery of the eye without rotating it. However, a competent and experienced assistant is not always available, and surgeons rarely feel safe if the eye is not totally in their own hands. Secondly, the usual 27 mm vitrector is not designed for pediatric eyes. When using a 27 mm adult vitrector in children's eyes, a surgeon has to hold the vitrector differently from the usual manner in adult vitrectomy, and the kid's nose more easily obstructs the surgeon's hands. Thirdly, the far-too-long probe might easily damage the macula or even the choroid with a slight slip of the hand.

The short vitrectomy kit is a great improvement in pediatric retinal surgeries. Currently, the available option is Alcon's short vitrectomy pak with a probe length of 18mm. Recently, DORC system also announced their Ultra-Short vitrectomy kit. They claim the 27-gauge short vitrector is 25% shorter and 60% stiffer than the usual-length 27-gauge vitrector, which makes its length around 20.25 mm. With an even shorter length at 18 mm, the Alcon's short vitrectomy probe possibly brings more efficacy and safety in surgery. The pediatric eyes are notoriously "non-forgiving" with iatrogenic retinal breaks. Due to this reason, surgeons tend to be more conservative in operating pediatric eyes, and if the surgery or instruments are not in perfect condition, they are prone to do very little and leave the eyes for a second surgery later on. The introduction of a shorter, stiffer probe might change this and help surgeons achieve better surgical goals and as well as better outcomes for the patient. However, the use of 18 mm short vitrector is very limited throughout the world, and there are no reports on single-arm outcomes or a comparative study using 18 mm versus 27 mm vitrector. Therefore, this study is proposed to gain more knowledge regarding the possible advantages of short vitrectomy for pediatric retinal surgeries.

Patients under 18 years of age who are scheduled for vitrectomy surgery due to various etiologies will be prospectively enrolled. Intraoperative complication rates, including lens injury and iatrogenic retinal breaks, will be recorded. The bending rate of the vitrector probe will be documented. A questionnaire regarding the overall comfort and confidence level of operating with a short vitrectomy will be filled out by the primary surgeon. Postoperatively, the ocular anatomical and functional outcomes and the rate of a second surgery will be documented. These data will be analyzed and compared with our previous pediatric vitrectomy cohort (using the 27 mm vitrectomy) to demonstrate the difference between the 18 mm and 27 mm probes.

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 18 years old
* Need vitrectomy due to various etiologies, including retinopathy of prematurity, familial exudative vitreoretinopathy, persistent fetal vasculature, congenital cataract, lens dislocation, open-globe injury, vitreous hemorrhage, or other vitreoretinal diseases.

Exclusion Criteria:

* Patients who cannot cooperate fully with detailed ophthalmic examinations.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
SAFETY of 18 mm vitrectomy probe in pediatric vitreoretinal surgery | Intraoperatively
  Incidence of iatrogenic injury as assessed by the percentage of surgery with iatrogenic injury event
SAFETY of 18 mm vitrectomy probe in pediatric vitreoretinal surgery | Intraoperatively
  Incidence of intraoperative instrument bending as assessed by the percentage of surgery with instrument bending event

SECONDARY OUTCOMES:
EFFICACY of 18 mm vitrectomy probe in pediatric vitreoretinal surgery | 6, 12, and 24 months postoperatively
  Incidence of retinal detachment as assessed by ophthalmoscopy
EFFICACY of 18 mm vitrectomy probe in pediatric vitreoretinal surgery | 6, 12, and 24 months postoperatively
  Visual acuity as assessed by the Snellen Chart
SATISFACTION of surgeon while using 18 mm short vitrectomy probe for pediatric vitreoretinal surgery | Intraoperatively
  The surgeon's satisfaction score as accessed by a satisfaction questionnaire that includes a scale from 0 (least satisfaction) to 5 (max satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Chi Wu, MD, PhD, Study Chair — Chang Gung Medical Foundation
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gan NY, Lam WC. Special considerations for pediatric vitreoretinal surgery. Taiwan J Ophthalmol. 2018 Oct-Dec;8(4):237-242. doi: 10.4103/tjo.tjo_83_18. PMID 30637195
- [Background] Yeh CT, Chen KJ, Liu L, Wang NK, Hwang YS, Chao AN, Chen TL, Lai CC, Wu WC. Visual and Anatomical Outcomes With Vitrectomy in Posterior or Combined Persistent Fetal Vasculature in an Asian Population. Ophthalmic Surg Lasers Imaging Retina. 2019 Jun 1;50(6):377-384. doi: 10.3928/23258160-20190605-06. PMID 31233155
- [Background] Huang YC, Chu YC, Wang NK, Lai CC, Chen KJ, Hwang YS, Wu WC. IMPACT OF ETIOLOGY ON THE OUTCOME OF PEDIATRIC RHEGMATOGENOUS RETINAL DETACHMENT. Retina. 2019 Jan;39(1):118-126. doi: 10.1097/IAE.0000000000001908. PMID 29190237
- [Background] Wang NK, Tsai CH, Chen YP, Yeung L, Wu WC, Chen TL, Lin KK, Lai CC. Pediatric rhegmatogenous retinal detachment in East Asians. Ophthalmology. 2005 Nov;112(11):1890-5. doi: 10.1016/j.ophtha.2005.06.019. PMID 16271317